CLINICAL TRIAL: NCT03580317
Title: Electroacupuncture Therapy for Change of Pain in Classical Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: Jiaxing TCM Hospital (Unknown)
Responsible Party: Principal Investigator, Jianqiao Fang, Professor, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018ZY008-CTN
Record Dates: First submitted 2018-06-02; First posted 2018-07-09 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Trigeminal Neuralgia
Keywords: Classical trigeminal neuralgia; Electroacupuncture; Randomized controlled clinical trial
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EA + Carbamazepine Group (Experimental): The subjects in this group will receive 3 times per week, and 4 weeks of continuous intervention for a total of 12 times. The intervention including electroacupuncture(EA) treatment and combined with Carbamazepine (0.1g each time, thrice daily). The follow-up period is 6 months.
  Interventions: Other: EA+ Carbamazepine
- EA + Placebo Group (Placebo Comparator): The subjects in this group will receive 3 times per week, and 4 weeks of continuous intervention for a total of 12 times. The intervention including EA treatment and combined with placebo of carbamazepine. The follow-up period is 6 months.
  Interventions: Other: EA+Placebo
- Sham EA+ Carbamazepine Group (Active Comparator): The subjects in this group will receive 3 times per week, and 4 weeks of continuous intervention for a total of 12 times. The intervention including sham electroacupuncture(sham EA) intervention and combined with carbamazepine. The follow-up period is 6 months.
  Interventions: Other: sham EA+Carbamazepine
- Sham EA+ Placebo Group (Sham Comparator): The subjects in this group will receive 3 times per week, and 4 weeks of continuous intervention for a total of 12 times. The intervention including sham EA intervention and combined with placebo took orally. The follow-up period is 6 months.
  Interventions: Other: sham EA+Placebo

INTERVENTIONS:
Other: EA+ Carbamazepine — Acupoints selection: Si-bai(ST2), Xia-guan(ST7), Di-cang(ST4), Quan-liao(SI18), Jia-che(ST6) and A-shi-xue of affected side. He-gu(LI4) and Wai-guan(TE5) of two sides.
  Operation:The needles(0.18×25 mm) will be selected to stimulate the local points with shallow row needling according to the distribution of neuropathy branch of trigeminal neuralgia.The needles(0.25×40mm) will be selected to stimulate the distal acupoints. The Xia-guan(ST7) and Quan-liao(SL18) (or Jia-che(ST6)), He-gu(LI4) and Wai-guan(SJ5) acupoints will be received EA treatment by HuaTuo SDZ-ⅡB acupoint neural stimulator. The EA parameter is 2/100 Hz, 60 minutes and the current intensity is comfortable to subjects. Carbamazepine tablets should be took orally, 0.1g each time, thrice daily.
  Arms: EA + Carbamazepine Group
Other: EA+Placebo — In this group, the selection, positioning and manipulation of acupoints, the frequency, duration and retaining needle time of treatment are same as EA + Carbamazepine Group; placebo, that appearance and specifications are the same as carbamazepine, are cooperated taken of dose 0.1g, thrice daily.
  Arms: EA + Placebo Group
Other: sham EA+Carbamazepine — Selection of points and locations: the non-meridional points which are means to the points beside 5-10mm of the real acupoints (avoid the trigger point) in the EA group will be selected and needled with more shallow acupuncture (the depth of needling is about 1-2mm).
  The operation of shame EA: The HuaTuo SDZ-ⅡB acupoint neural stimulator with damaged electrode wires will be selected to connect the points next to the Xia-guan(ST7) and Quan-liao (SI18) , He-gu (LI4) and Wai-guan(TE5).The frequency, intensity and retaining time will be same as EA group, The subjects can see the display screen and parameter settings of stimulator, however there is no electricity output in fact.
  The dosage and frequency of oral carbamazepine tablets are same as above part.
  Arms: Sham EA+ Carbamazepine Group
Other: sham EA+Placebo — The points selection, positioning and manipulation are same as Shame EA+ Carbamazepine group，placebo are cooperated taken of dose 0.1g, thrice daily.
  Arms: Sham EA+ Placebo Group

SUMMARY:
The classical trigeminal neuralgia (CTN) is a common neuropathic pain in clinic by recurrent attacks of chronic sharp pain in the distribution of neuropathy branches of trigeminal neuralgia. With the lack of appropriate drug and surgery, acupuncture played a role in analgesia with its effective and few side effects. The study is designed to observe the therapeutic effect and safety of electroacupuncture (EA) in the treatment of CTN.

DETAILED DESCRIPTION:
A total of 120 subjects with CTN who met the inclusion criteria will be included in the study. The subjects will be randomly divided into EA+ Carbamazepine group, EA+placebo group, sham EA+Carbamazepine group and sham EA+placebo group. The indexes of main outcome evaluation are 1)Intensity of pain (Evaluation of the pain by VAS with 0-10 points) and 2)Brief introduction of 2-week pain. The indexes of secondary outcome evaluation are 1) Brief Pain Inventory-Facial scale(BPI-Facial); 2) Patient Global Impression of Change(PGIC); 3) Short-Form McGill Pain Questionnaire; 4) Short- Form 36 Questionnaire. This study will evaluate whether EA has the advantage over carbamazepine in the immediate effect, long-term effect and post effect of the analgesia in CTN. At the same time, the study also will demonstrate whether EA has a synergistic effect with carbamazepine on the treatment of CTN, or even whether EA has an alternative effect on carbamazepine. Furthermore, we will establish a standardized, effective and convenient therapy program of EA to promote according to the results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffer from the pain with electric shock, shooting, stabbing occurs in one or more branches of the trigeminal nerve.
2. The visual analogue score(VAS) baseline score ≥5, have a attack more than 3 times a day, at least 4 days a week.
3. 18 years ≤ age ≤ 80 years.
4. Clear consciousness, have the ability of pain perception and resolution, can complete the basic communication.
5. Signed informed consent and volunteered to participate in this study.

Exclusion Criteria:

1. Those patients with epilepsy, head injury or other related neurological diseases.
2. Patients with serious heart, liver, kidney damage or cognitive impairment, aphasia, mental disorders, or unable to cooperate with the treatment.
3. Combined with hypertension but poor control.
4. Severe depressive with definitive diagnosis recently.
5. Pregnant and lactating patients.
6. Installing pacemakers.
7. For any other reason that is not suitable for the treatment of EA.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Intensity of Pain to 28 weeks | Baseline, 2 weeks, 4 weeks, 16 weeks, 28 weeks
  Evaluation of the pain by VAS with 0-10 points which that 0 means painless and 10 means very painful.

SECONDARY OUTCOMES:
Brief Pain Inventory-Facial scale(BPI-Facial) | Baseline, 2 weeks, 4 weeks, 16 weeks, 28 weeks
  This instrument is composed of 18 items on a 1-point scale (0-10). 4 questions center on pain intensity, 7 questions deal with the interference of pain with general life activities and the remaining 7 questions deal with the interference of pain with face-specific activities.
Patient Global Impression of Change(PGIC) | Baseline, 2 weeks, 4 weeks, 16 weeks, 28 weeks
  This index will record the general change impression of pain for CTN.
Short-Form McGill Pain Questionnaire | Baseline, 2 weeks, 4 weeks, 16 weeks, 28 weeks
  The pain rating index has 2 subscales: these words or items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe. There's also one item for present pain intensity and one item for a 10cm visual analogue scale for average pain. This version includes 7 additional symptoms related to neuropathic pain, for a total of 22 items with 0-10 numerical response options.
Short-Form 36 Questionnaire | Baseline, 2 weeks, 4 weeks, 16 weeks, 28 weeks
  The scale includes: 1.Physical Functioning (PF).2.Physical function (RP).3.Body Pain (BP).4.General Health (GH).5.Vitality.6.Social Functioning (SF)7.Role-emotional (RE).8.Mental Health (MH).
The proportion of patients using rescue analgesics | Baseline, 2 weeks, 4 weeks, 16 weeks, 28 weeks
  The proportion of patients using rescue analgesics
The frequency of CTN attacks | Baseline, 2 weeks, 4 weeks, 16 weeks, 28 weeks
  Calculated from the pain diary

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D,M.D, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montano N, Conforti G, Di Bonaventura R, Meglio M, Fernandez E, Papacci F. Advances in diagnosis and treatment of trigeminal neuralgia. Ther Clin Risk Manag. 2015 Feb 24;11:289-99. doi: 10.2147/TCRM.S37592. eCollection 2015. PMID 25750533
- [Background] van Kleef M, van Genderen WE, Narouze S, Nurmikko TJ, van Zundert J, Geurts JW, Mekhail N; World Institute of Medicine. 1. Trigeminal neuralgia. Pain Pract. 2009 Jul-Aug;9(4):252-9. doi: 10.1111/j.1533-2500.2009.00298.x. PMID 19619267
- [Background] Wiffen PJ, Derry S, Moore RA, Kalso EA. Carbamazepine for chronic neuropathic pain and fibromyalgia in adults. Cochrane Database Syst Rev. 2014 Apr 10;2014(4):CD005451. doi: 10.1002/14651858.CD005451.pub3. PMID 24719027
- [Background] Killian JM, Fromm GH. Carbamazepine in the treatment of neuralgia. Use of side effects. Arch Neurol. 1968 Aug;19(2):129-36. doi: 10.1001/archneur.1968.00480020015001. No abstract available. PMID 4877400
- [Background] Wiffen PJ, McQuay HJ, Moore RA. Carbamazepine for acute and chronic pain. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD005451. doi: 10.1002/14651858.CD005451. PMID 16034977
- [Background] Zhang R, Lao L, Ren K, Berman BM. Mechanisms of acupuncture-electroacupuncture on persistent pain. Anesthesiology. 2014 Feb;120(2):482-503. doi: 10.1097/ALN.0000000000000101. PMID 24322588
- [Background] Wu CH, Lv ZT, Zhao Y, Gao Y, Li JQ, Gao F, Meng XF, Tian B, Shi J, Pan HL, Li M. Electroacupuncture improves thermal and mechanical sensitivities in a rat model of postherpetic neuralgia. Mol Pain. 2013 Apr 3;9:18. doi: 10.1186/1744-8069-9-18. PMID 23551937
- [Background] Aranha MF, Muller CE, Gaviao MB. Pain intensity and cervical range of motion in women with myofascial pain treated with acupuncture and electroacupuncture: a double-blinded, randomized clinical trial. Braz J Phys Ther. 2015 Jan-Feb;19(1):34-43. doi: 10.1590/bjpt-rbf.2014.0066. Epub 2014 Nov 28. PMID 25714602
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299
- [Background] Truini A, Galeotti F, Cruccu G. New insight into trigeminal neuralgia. J Headache Pain. 2005 Sep;6(4):237-9. doi: 10.1007/s10194-005-0195-9. PMID 16362674
- [Background] Cruccu G, Biasiotta A, Galeotti F, Iannetti GD, Innocenti P, Romaniello A, Truini A. Diagnosis of trigeminal neuralgia: a new appraisal based on clinical and neurophysiological findings. Suppl Clin Neurophysiol. 2006;58:171-86. doi: 10.1016/s1567-424x(09)70067-4. No abstract available. PMID 16623330
- [Background] Chen GQ, Wang XS, Wang L, Zheng JP. Arterial compression of nerve is the primary cause of trigeminal neuralgia. Neurol Sci. 2014 Jan;35(1):61-6. doi: 10.1007/s10072-013-1518-2. Epub 2013 Aug 21. PMID 23963805
- [Background] Jia DZ, Li G. Bioresonance hypothesis: a new mechanism on the pathogenesis of trigeminal neuralgia. Med Hypotheses. 2010 Mar;74(3):505-7. doi: 10.1016/j.mehy.2009.09.056. Epub 2009 Nov 8. PMID 19900765
- [Background] Devor M, Amir R, Rappaport ZH. Pathophysiology of trigeminal neuralgia: the ignition hypothesis. Clin J Pain. 2002 Jan-Feb;18(1):4-13. doi: 10.1097/00002508-200201000-00002. PMID 11803297
- [Background] Zakrzewska JM, Linskey ME. Trigeminal neuralgia. BMJ. 2014 Feb 17;348:g474. doi: 10.1136/bmj.g474. No abstract available. PMID 24534115
- [Derived] Li R, Sun J, Luo K, Luo N, Sun R, Gao F, Wang Y, Xia Y, Li X, Chen L, Ma R, Shao X, Liang Y, Fang J. Electroacupuncture and carbamazepine for patients with trigeminal neuralgia: a randomized, controlled, 2 x 2 factorial trial. J Neurol. 2024 Aug;271(8):5122-5136. doi: 10.1007/s00415-024-12433-x. Epub 2024 May 31. PMID 38816482

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03580317/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03580317/ICF_001.pdf